CLINICAL TRIAL: NCT05955014
Title: Data Collection Protocol for Patients With Von Hippel Lindau Disease
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0665; NCI-2023-05216 (Other: NCI-Clinical Trials Registry)
Record Dates: First submitted 2023-07-10; First posted 2023-07-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Von Hippel Lindau Disease
MeSH Terms: conditions — von Hippel-Lindau Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To collect information from patients with vHL disease. Information collected will include data on the status of the disease, any surgeries or therapies patients have received for vHL disease, and quality of life.

DETAILED DESCRIPTION:
Primary Objectives:

* Obtain prospective and retrospective data on lesion development, surgical history and systemic therapy use in patients with vHL disease
* Assess genotype-phenotype correlation between VHL mutation type and patterns of lesion development
* Assess genotype-phenotype correlation for response to belzutifan in an organ-specific manner

Secondary Objectives:

--Obtain quality of life data in patients with vHL disease

ELIGIBILITY:
Inclusion Criteria:

* Presence of genetic confirmation or clinical criteria consistent with vHL disease.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

• Patients with psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: M D Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jonasch, MD, Principal Investigator — ejonasch@mdanderson.org
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org